CLINICAL TRIAL: NCT04695951
Title: Efficacy and Safety of Renalof® in the Removal of Calculi Smaller Than 10 mm Located in the Reno-Ureteral Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201920-RENALOF-NI
Record Dates: First submitted 2020-12-15; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Renal Injury; Kidney Injury; Kidney Calculi; Ureteral Obstruction; Ureteral Calculi; Renal Stone; Ureteral Injury; Renal Disease; Urolithiasis, Calcium Oxalate; Urolithiasis; Lower Urinary Tract; Urolithiasis
Keywords: Urolithiasis; Kidney Stone; Agropyron Repens; Ureteral calculi; Calcium oxalate
MeSH Terms: conditions — Kidney Calculi; Ureteral Obstruction; Ureteral Calculi; Nephrolithiasis; Kidney Diseases; Nephrolithiasis, Calcium Oxalate; Urolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renalof (Experimental): A total of 120 patients treated with the study product Renalof® at a dose of 650 mg twice daily were followed for 4 months. A preliminary analysis of the types of stones present in the study patients was performed according to the main compound, using a biophysical profile by biochemical analysis and the clinical characteristics, medical history and biochemical profile of the creatinine values of the test patients. Imaging and quality of life tests were carried out during the trial to check the efficacy and possible adverse effects of the test product in patients with kidney stones.
  Interventions: Dietary Supplement: Renalof
- Control (Placebo Comparator): A total of 35 patients treated with the study product Placebo at a dose of 650 mg twice daily were followed for 4 months. A preliminary analysis of the types of stones present in the study patients was performed according to the main compound, using a biophysical profile by biochemical analysis and the clinical characteristics, medical history and biochemical profile of the creatinine values of the test patients. Imaging and quality of life tests were carried out during the trial to check the efficacy and possible adverse effects of the test product in patients with kidney stones.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Renalof — A total of 120 patients treated with the study product Renalof® at a dose of 650 mg twice daily were followed for 4 months. A preliminary analysis of the types of stones present in the study patients was performed according to the main compound, using a biophysical profile by biochemical analysis and the clinical characteristics, medical history and biochemical profile of the creatinine values of the test patients. Imaging and quality of life tests were carried out during the trial to check the efficacy and possible adverse effects of the test product in patients with kidney stones.
  Arms: Renalof
Other: Placebo — A total of 35 patients treated with Placebo at a dose of 650 mg twice daily were followed for 4 months. A preliminary analysis of the types of stones present in the study patients was performed according to the main compound, using a biophysical profile by biochemical analysis and the clinical characteristics, medical history and biochemical profile of the creatinine values of the test patients. Imaging and quality of life tests were carried out during the trial to check the efficacy and possible adverse effects of the test product in patients with kidney stones.
  Arms: Control

SUMMARY:
Given the high recurrence of urolithiasis in patients, the search for less aggressive and preventive treatments is increasingly necessary. Renalof® is presented as an alternative to herbal medicine being a product that, due to its diuretic and demineralization properties of kidney stones, has been widely used in this patient population, disintegrating and eliminating calcium oxalate and struvite stones in a painless in the genitourinary system.

With the objective of determining the efficacy of this therapy, an observational, prospective, randomized, single-blind, two-arm study was carried out: treatment group with Renalof® and control group, placebo.

DETAILED DESCRIPTION:
Given the high recurrence of urolithiasis in patients, the search for less aggressive and preventive treatments is increasingly necessary. Renalof® is presented as an alternative to herbal medicine being a product that, due to its diuretic and demineralization properties of kidney stones, has been widely used in this patient population, disintegrating and eliminating calcium oxalate and struvite stones in a painless in the genitourinary system.

With the objective of determining the efficacy of this therapy, an observational, prospective, randomized, single-blind, two-arm study was carried out: treatment group with Renalof® and control group, placebo.

The treatment group consists of 120 patients over 18 years of age, of both sexes, with a diagnosis of urolithiasis less than 10 mm in diameter, present throughout the entire reno-uretero-bladder path, diagnosed by ultrasound, renal CT and urography . The Renalof® product was administered at a dose of 650 mg daily for 3 months and the presence of stones in any location of the reno-ureteral tract was evaluated using one of the diagnostic means mentioned in monthly consultations. The second group, treated with placebo corresponding to 35 people constituting 30% of the universe. The study period was from August 2019 to July 2020 at the Hospital Escuela Antonio Lenin Fonseca and the Seniors clinic, in the city of Managua, Nicaragua.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years of age, in all their mental and physical capacities to decide to be part of this study.
2. There are no comorbidities or associated diseases that put the stability of the patient at risk.
3. Not be diagnosed as Chronic Kidney Disease, in any stage.
4. Existence of non-obstructive stones smaller than 10 mm located in the renoureteral path.
5. No compromise of renal viability.

Exclusion Criteria:

1. Patients under 18 years of age.
2. Existence of comorbidities or associated diseases that put the stability of the patient at risk.
3. Existence of a diagnosis of Chronic Kidney Disease, at any stage.
4. Presence of non-obstructive or obstructive stones greater than 10 mm located in the renoureteral path.
5. Renal viability compromise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
kidney stone clearance with Renalof® treatment compared to placebo | 4 months
  kidney stone clearance with Renalof® treatment compared to placebo measured by ultrasound and tomography imaging

SECONDARY OUTCOMES:
Quality of life of patients | 4 months
  Quality of life was established in relation to the presence or absence of symptoms related to the disease by means of a bimonthly personal questionnaire: dysuria or burning when urinating, urinary urgency, kidney colic, difficulty in performing daily activities and periodicity of urinary infections (mild, moderate, severe, yes or no,).
Number of colic | 4 months
  number of colic during the 4-month follow-up of treatment
Adverse events related with product of the trial | 4 months
  Adverse effects related with the test product in patients with kidney stones, measured by means of a bimonthly personal questionnaire: nausea, vomiting, digestive pain, stomach ache... (mild, moderate, severe, yes or no,).

OTHER OUTCOMES:
Cost of treatment | 4 months
  cost of treatment with the use of Renalof® compared to the usual treatments, taking into account hospitalization time due to the number of colic and recovery time due to urolithiasis

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Seniors Managua, Managua, Nicaragua

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Tsujihata M. Mechanism of calcium oxalate renal stone formation and renal tubular cell injury. Int J Urol. 2008 Feb;15(2):115-20. doi: 10.1111/j.1442-2042.2007.01953.x. PMID 18269444
- [Background] Johnson CM, Wilson DM, O'Fallon WM, Malek RS, Kurland LT. Renal stone epidemiology: a 25-year study in Rochester, Minnesota. Kidney Int. 1979 Nov;16(5):624-31. doi: 10.1038/ki.1979.173. PMID 548606
- [Background] Soucie JM, Coates RJ, McClellan W, Austin H, Thun M. Relation between geographic variability in kidney stones prevalence and risk factors for stones. Am J Epidemiol. 1996 Mar 1;143(5):487-95. doi: 10.1093/oxfordjournals.aje.a008769. PMID 8610664
- [Background] Wesson JA, Johnson RJ, Mazzali M, Beshensky AM, Stietz S, Giachelli C, Liaw L, Alpers CE, Couser WG, Kleinman JG, Hughes J. Osteopontin is a critical inhibitor of calcium oxalate crystal formation and retention in renal tubules. J Am Soc Nephrol. 2003 Jan;14(1):139-47. doi: 10.1097/01.asn.0000040593.93815.9d. PMID 12506146
- [Background] Kohri K, Yasui T, Okada A, Hirose M, Hamamoto S, Fujii Y, Niimi K, Taguchi K. Biomolecular mechanism of urinary stone formation involving osteopontin. Urol Res. 2012 Dec;40(6):623-37. doi: 10.1007/s00240-012-0514-y. Epub 2012 Nov 6. PMID 23124115
- [Background] Mykoniatis I, Sarafidis P, Memmos D, Anastasiadis A, Dimitriadis G, Hatzichristou D. Are endourological procedures for nephrolithiasis treatment associated with renal injury? A review of potential mechanisms and novel diagnostic indexes. Clin Kidney J. 2020 May 22;13(4):531-541. doi: 10.1093/ckj/sfaa020. eCollection 2020 Aug. PMID 32905259
- [Background] Grases F, Ramis M, Costa-Bauza A, March JG. Effect of Herniaria hirsuta and Agropyron repens on calcium oxalate urolithiasis risk in rats. J Ethnopharmacol. 1995 Mar;45(3):211-4. doi: 10.1016/0378-8741(94)01218-o. PMID 7623486
- [Background] Beydokthi SS, Sendker J, Brandt S, Hensel A. Traditionally used medicinal plants against uncomplicated urinary tract infections: Hexadecyl coumaric acid ester from the rhizomes of Agropyron repens (L.) P. Beauv. with antiadhesive activity against uropathogenic E. coli. Fitoterapia. 2017 Mar;117:22-27. doi: 10.1016/j.fitote.2016.12.010. Epub 2016 Dec 29. PMID 28040531
- [Background] Paslawska S, Piekos R. Studies on the optimum conditions of extraction of silicon species from plants with water. IV. Agropyron repens. Planta Med. 1976 Nov;30(3):216-22. doi: 10.1055/s-0028-1097720. No abstract available. PMID 1005521
- [Background] Bragadottir G, Redfors B, Ricksten SE. Mannitol increases renal blood flow and maintains filtration fraction and oxygenation in postoperative acute kidney injury: a prospective interventional study. Crit Care. 2012 Aug 17;16(4):R159. doi: 10.1186/cc11480. PMID 22901953
- [Background] Hagerstrom E, Lindberg L, Bentzen J, Brodbaek K, Zerahn B, Kristensen B. The Nephroprotective Effect of Mannitol in Head and Neck Cancer Patients Receiving Cisplatin Therapy. Clin Med Insights Oncol. 2019 Jan 7;13:1179554918821320. doi: 10.1177/1179554918821320. eCollection 2019. PMID 30670924